CLINICAL TRIAL: NCT01156623
Title: Value of EBUS-TBNA for Mediastinal Lymph Nodes in Non-small Cell Lung Cancer in a Tuberculosis-endemic Country
Brief Title: Endobronchial Ultrasound Guided Transbronchial Aspiration (EBUS-TBNA) in Non Small Cell Lung Cancer (NSCLC) in a Tuberculosis-endemic Country
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung Fu-Tsai, Attending physician, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 98-3639A3
Record Dates: First submitted 2010-06-30; First posted 2010-07-05 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EBUS-TBNA; NSCLC; Mediastinal lymph node; tuberculosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With EBUS-TBNA group (Experimental): The patients enrolled in present study are those with non-small lung cancer and receive contrast-enhanced computed tomography (CT) and Positron emission tomography (PET) with fluorine-18 fluorodeoxyglucose (FDG) examination. In this group, further EBUS-TBNA will be arranged if patients agreed it.
  Interventions: Procedure: EBUS-TBNA
- Without EBUS-TBNA group (No Intervention): The patients enrolled in present study are those with non-small lung cancer and receive contrast-enhanced computed tomography (CT) and Positron emission tomography (PET) with fluorine-18 fluorodeoxyglucose (FDG) examination. In this group, no EBUS-TBNA will be arranged if patients refused it despite we advised it.

INTERVENTIONS:
Procedure: EBUS-TBNA — All included patients received TBNA for lymph node study via a flexible ultrasonic bronchoscope with a linear scanning probe on the tip (BF-UC206F-OL8, Olympus). The curved-probe scanned parallel to the insertion direction of bronchoscope, and the obtained images were linked to the ultrasound scanner (EU-2000C, Olympus) incorporated with Doppler-flow imaging. Each lymph node greater than 5mm in short axis measured by cursors was selected for subsequent TBNA with a 22-gauge (NA-201SX-4022, Olympus) needle in a condition of real-time EBUS guidance. A cytology examination was sent for pathologist blinded for the clinical history and image result of patients. When a tissue core was obtained by TBNA, the specimen was also sent for pathology study.
  Arms: With EBUS-TBNA group

SUMMARY:
In lung cancer with enlarged or non-enlarged mediastinal lymph nodes, contrast-enhanced computed tomography (CT) and Positron emission tomography (PET) scan frequently show discrepancy in tuberculosis-endemic area. Endobronchial ultrasound guided transbronchial aspiration (EBUS-TBNA) with ability of real-time nodal sampling possibly improves the nodal diagnosis.

The purpose of this study is to compare the accuracy of nodal diagnosis of contrast-enhanced CT and PET scan with and without EBUS-TBNA, this study will be performed.

DETAILED DESCRIPTION:
Lung cancer remains a fatal disease worldwide, and surgical treatment offers possibility for long-term survival. However, the indication and outcome of surgical resection depends on the pre-operative accurate staging and extent of intra-operative lymph node dissection. Therefore, the accurate lymph node staging in non-small cell lung cancer (NSCLC) is crucial for planning optimal treatment. Traditionally, the conventional contrast-enhanced CT essentially identifies enlarged lymph node greater than 1cm as nodal metastasis. Nevertheless, with moderate sensitivity and specificity, contrast-enhanced CT carries substantial risk to under-stage small nodal metastasis and to over-stage inflammatory lymphadenitis.

Positron emission tomography (PET) with fluorine-18 fluorodeoxyglucose (FDG) provides functional images of tumor metabolism, and has been used as a non-invasive alternative other than contrast-enhanced CT for nodal staging in NSCLC. In the absence of detectable lymph node enlargement by CT, FDG-PET scan were increasingly used to stage the lymph node status for NSCLC in some part of world. Hence, the accuracy of FDG-PET might substantially alter the treatment strategy in an institution where the mediastinoscopy is unavailable for lymph node sampling. However, it is generally agreed that abnormal FDG uptake occurred frequently in granulomatous and inflammatory disease. In an endemic area where tuberculosis is still prevalent; such as Eastern Asia, FDG-PET scan has reportedly shown reduced sensitivity and positive predictive value in nodal staging of NSCLC. Thereby, FDG-PET scan alone does not appear to replace mediastinoscopy for nodal staging of NSCLC in a tuberculosis-endemic area, especially in potentially operable patients without enlarged mediastinal lymph nodes.

The recent development of curved ultrasound probe-equipped bronchoscope, which enables direct and real-time aspiration by endobronchial ultrasound- transbronchial needle aspiration (EBUS-TBNA) of mediastinal and hilar lymph nodes, has become an less invasive alternative for nodal staging other than mediastinoscopy. By direct nodal sampling, EBUS-TBNA improves lymph node staging from an image basis to a cytology basis; or even, pathology basis. However, the variable sensitivity and negative predictive value of EBUS-TBNA has been reported, especially in lymph node reduced in size after induction chemotherapy. Nevertheless, reports from NSCLC without significant mediastinal lymph node enlargement on CT otherwise suggested EBUS-TBNA exhibited a high sensitivity and specificity for detecting small nodal metastasis. Therefore, whether EBUS-TBNA retains the reportedly high performance of nodal staging in lung cancer patients without enlarged mediastinal lymph node on CT in a TB endemic country; a condition of FDG-PET scan reportedly showed increased false-positive rate, is still unclear.

In present study, we primarily aim at the comparison of accuracy of nodal diagnosis of contrast-enhanced CT and PET scan with and without EBUS-TBNA in a condition of mediastinal and hilar lymph nodes of lung cancer. Secondarily, we aim at the accuracy of nodal diagnosis by FDG-PET scan in the same condition, and investigate the characteristics of lymph nodes with false PET result.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC,
* Completed whole body CT or PET scan.

Exclusion Criteria:

* Pregnancy,
* Age less than 20 years old,
* Other malignancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2012-10 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 2 weeks
  The results of each diagnostic modality were compared with the surgical pathology obtained by thoracotomy and lymph node dissection. The sensitivity, specificity, positive predictive value and negative predictive value of each diagnostic modality were calculated as the standard definition.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tsai Chung, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taipei, Taiwan